CLINICAL TRIAL: NCT00951964
Title: Treatment of Epidermolysis Bullosa Dystrophica by Polyphenon E (Epigallocatechin 3 Gallate)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 09-APN-01
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): patients receive the treatment in first and placebo in second part of study
  Interventions: Drug: Polyphenon E before Placebo
- 2 (Other): patients receive placebo in first and treatment in second part of study
  Interventions: Drug: placebo before treatment

INTERVENTIONS:
Drug: Polyphenon E before Placebo — patients receive polyphenon E during 4 months, then 2 months of wash-out and finally 4 months of placebo
  Arms: 1
Drug: placebo before treatment — patients receive 4 months of placebo, then 2 months of wash out et finally 4 months of treatment
  Arms: 2

SUMMARY:
Dystrophic epidermolysis bullosa hereditaria are genodermatosis responsible for formation of cutaneous bullous lesion arising spontaneously or after mechanical trauma.

These lesions are due to mutation on gene COL7A1 coding for collagen VII. There is no treatment available. Cares are consisting to dress lesions and to protect the skin.

The investigators have recently observed on patients having residual expression of collagen VII that phenotype severity is modulated by activation degree of dermic metalloproteinase. The investigators have also observed that epigallocatechin-3-gallate (Polyphenon E®) could be regulated this activity.

The primary purpose of this study is to assessing the efficacity of Polyphenon E to decrease the number of cutaneous bullosa after four month of treatment.

The primary outcome measure is the rate of patient presenting a decrease of 20% or more of the number of cutaneous bullosa.

Secondary outcomes are: severity of mucosa impairment, affected cutaneous surface, the average duration of cicatrisation and treatment tolerance.

This study foresees the inclusion of 22 patients older than 2 years old in 5 centers.

When patients are included, they will be randomized and receive the treatment (or placebo) for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* known mutation of COL7A1

Exclusion Criteria:

* tea drinkers
* patient receiving induction treatment,protease inhibitor treatment
* liver failure

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
decrease of number of cutaneous bullosa | after 4 months of treatment

SECONDARY OUTCOMES:
efficacity of treatment | at 4 , 6, 7 10 months after beginnig of treatment and at year 1
tolerance tio treatment | at 1, 4, 6, 7, 10 and 12 months after beginnig the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chiaverini, PhD, Principal Investigator — dermatology department, Nice University Hospital
Locations (5):
- France (5):
  - Dermatology Department, Bordeaux University Hospital, Bordeaux
  - Dijon University Hospital, Dermatology Department, Dijon
  - Dermatology Department, Necker Enfants Malades, APHP, Paris
  - Dermatology Department, Saint Louis Hospital, APHP, Paris
  - Toulouse University Hospital, Dermatology Department, Toulouse

REFERENCES:
- [Derived] Chiaverini C, Roger C, Fontas E, Bourrat E, Bourdon-Lanoy E, Labreze C, Mazereeuw J, Vabres P, Bodemer C, Lacour JP. Oral epigallocatechin-3-gallate for treatment of dystrophic epidermolysis bullosa: a multicentre, randomized, crossover, double-blind, placebo-controlled clinical trial. Orphanet J Rare Dis. 2016 Mar 25;11:31. doi: 10.1186/s13023-016-0411-5. PMID 27015660